CLINICAL TRIAL: NCT04857476
Title: Do Patients With Skin PSoriasis Have Sub-clinical Features of ACTive Psoriatic Arthritis on Musculoskeletal UltraSound?
Acronym: PsACT-US
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to work commitment and time constraints, the study had to finish early..
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021RHE115
Record Dates: First submitted 2021-04-21; First posted 2021-04-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- skin psoriasis participants (Other): Single arm study
  Interventions: Diagnostic Test: Ultrasound scan

INTERVENTIONS:
Diagnostic Test: Ultrasound scan — Psoriasis epidemiology screening tool (PEST) score for completion Brief questionnaire about current psoriasis symptoms, current treatment and if any features associated with psoriatic arthritis.
  One-off musculo-skeletal ultrasound Questionnaire at 2 years

SUMMARY:
Psoriatic Arthritis is an inflammatory condition that typically affects joints and soft tissues such as tendons. Poorly controlled or untreated psoriatic arthritis can lead to joint damage, disability and poor physical and mental wellbeing. Evidence suggests that early diagnosis and treatment of psoriatic arthritis can minimise adverse health outcomes.

Musculoskeletal ultrasound has become an extremely useful tool in aiding rheumatologists to diagnose inflammatory joint conditions particularly at an early stage in the course of a disease.

Psoriatic arthritis is known to affect up to 30% of patients with skin psoriasis. Therefore, national dermatology guidelines advise that patients with skin psoriasis should be asked about any joint symptoms at least every year.

This study investigates whether skin psoriasis patients who are not on biologic treatment are indeed being asked about any joint symptoms and we subsequently invite patients for a musculoskeletal ultrasound scan to see if they have features of early psoriatic arthritis on ultrasound. Those who do are then invited for a thorough rheumatology clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Psoriasis by a dermatologist
* Aged 18 or more
* Reasonable fluency of spoken English

Exclusion Criteria:

* Existing diagnosis of Psoriatic arthritis
* Currently on biologics for treatment of their skin Psoriasis (as this would potentially treat and thereby diminish joint symptoms associated with PsA)
* Aged <18years old (the study focusses on an adult population)
* Currently in prison (would be unable to attend the study ultrasound scan)
* Unable to give written consent for a musculoskeletal ultrasound e.g. advanced dementia, learning difficulties (may be unable to appreciate the reason for the study and may be unable to tolerate sitting relatively still for an ultrasound scan for 60 minutes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with known skin psoriasis have features in keeping with psoriatic arthritis on musculoskeletal ultrasound | 3 years
  proportion of patients with known skin psoriasis have features in keeping with psoriatic arthritis on musculoskeletal ultrasound
Risk factors associated with those psoriasis patients who do have features of psoriatic arthritis on musculoskeletal ultrasound | 3 years
  Are there any particular risk factors associated with those psoriasis patients who do have features of psoriatic arthritis on musculoskeletal ultrasound?
PEST Scores | 3 years
  To identify whether patients who have higher PEST scores are more likely to have features of psoriatic arthritis on ultrasound
PEST score element | 3 years
  Which element of a PEST score, if reported by a patient, is most likely to be associated with features of psoriatic arthritis on musculoskeletal ultrasound
High PEST score with normal ultrasound scan | 2 years
  Are patients with a high PEST score and a normal initial musculoskeletal ultrasound scan more likely to be diagnosed with Psoriatic arthritis after 2 years

CONTACTS AND LOCATIONS:
Overall Officials: George Hirsch, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- George Hirsch, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No